CLINICAL TRIAL: NCT05163548
Title: Early Feasibility Study of the Vivasure PerQseal®+ (PerQseal® Plus) Vascular Closure Device When Used to Achieve Hemostasis of Common Femoral Arteriotomies Created by 14 to 22 F Sheaths in Patients Undergoing Percutaneous Transcatheter Procedures
Brief Title: PerQseal®+ Early Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivasure Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P856-00
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Percutaneous Large Hole Vascular Closure
Keywords: vascular closure; vascular closure device; large hole percutaneous closure; large bore percutaneous closure
MeSH Terms: interventions — Vascular Closure Devices

STUDY DESIGN:
Intervention Model Description: Early Feasibility Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Subjects that receive PerQseal Plus Device (Experimental): Subjects undergoing large hole endovascular percutaneous procedures with a femoral arteriotomy created with 14 to 22 F sheaths (arteriotomy up to 26 F)
  Interventions: Device: PerQseal Plus Device

INTERVENTIONS:
Device: PerQseal Plus Device — Percutaneous closure of femoral artery access site created by 14 to 22 F sheaths (up to 26 F arteriotomy) in patients undergoing Percutaneous Transcatheter procedures.
  Other Names: Vascular Closure Device

SUMMARY:
The objective of this Early Feasibility Study (EFS) is to evaluate the initial safety and preliminary effectiveness of the PerQseal®+ VCD in a small number of subjects when used to achieve hemostasis of common femoral arteriotomies created by 14 to 22 F sheaths (arteriotomy up to 26 F) in subjects undergoing Percutaneous Transcatheter procedures.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, single arm EFS. Patients undergoing a percutaneous trancatheter procedure, requiring an arteriotomy created by 14 - 22 F sheaths (arteriotomies up to approx. 26 F), via the common femoral artery will be screened against the study inclusion/exclusion criteria. If the patient meets study eligibility requirements, they shall be invited to participate, provide informed consent, and shall subsequently be assigned a study ID number. Enrollment will occur at the point where the PerQseal®+ VCD study device first enters the patient's body.

The planned enrollment is 15 treated patients at a maximum of 5 study sites (minimum of 3) located in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years, 2. Clinically indicated for a large bore interventional transcatheter procedure, e.g., transcatheter aortic valve repair (TAVR) or endovascular abdominal aortic aneurysm repair (EVAR), or thoracic endovascular aneurysm repair (TEVAR) using a percutaneous common femoral arteriotomy created by a 14 to 22 F sheath, 3. Subject is willing and able to provide appropriate study-specific informed consent, follow protocol procedures, and comply with follow-up visit requirements, 4. Females who are not pregnant or lactating and not planning to become pregnant for the duration of the study.

-

Exclusion Criteria:

Baseline Exclusion Criteria 1. Evidence of systemic bacterial or cutaneous infection, including groin infection Baseline Exclusion Criteria

1. Evidence of systemic bacterial or cutaneous infection, including groin infection,
2. Known bleeding diathesis, definite or potential coagulopathy, platelet count < 100,000/µl or subjects on long term anticoagulants with an INR > 2 within 12 hours prior to index procedure,
3. Significant anemia (hemoglobin < 9 g/dL or hematocrit < 27%), within 24 hours prior to index procedure,
4. Known type II heparin-induced thrombocytopenia,
5. NYHA functional class IV heart failure that is uncontrolled and requires treatment in the Intensive Care Unit, within 24 hours prior to primary procedure,
6. Documented left ventricular ejection fraction < 20%,
7. Unilateral or bilateral lower extremity amputation.
8. Claudication (e.g., Rutherford category 3 or greater), documented untreated iliac or common femoral artery diameter stenosis > 50% or previous bypass surgery/stent placement in the common femoral artery of target leg,
9. Known existing nerve damage in the target leg,
10. Renal insufficiency (Glomerular Filtration Rate ≤ 30 ml/min or baseline serum creatinine > 2.5 mg/dL) or on renal replacement therapy,
11. Known allergy to any of the materials used in the PerQseal®+ device (refer to Instructions for Use),
12. Subject unsuitable for surgical repair of the target leg access site,
13. Subject has undergone a percutaneous procedure greater than 8 F sheath in the target leg, within the 90 days prior to index procedure,
14. Subject has undergone use of an intra-aortic balloon pump through the target leg access site within 90 days prior to the index procedure,
15. Subject has undergone a percutaneous procedure of 8 F sheath or less using an absorbable intravascular closure device for hemostasis, in the target vessel, within the 90 days prior to index procedure,
16. Subject has undergone a percutaneous procedure of 8 F sheath or less using a suture mediated closure device or manual/mechanical pressure for hemostasis in the target leg, within the 30 days prior to index procedure,
17. Evidence of marked tortuosity of the femoral or external iliac artery in the target leg, based on pre-primary procedure CT angiography,
18. Evidence of arterial diameter stenosis > 30% within 15 mm proximal or distal to arteriotomy site based on pre-primary procedure CT angiography,
19. Evidence of anterior wall calcification of the target common femoral artery (other than small, diffuse deposits which in the opinion of the investigator will not impede the vascular closure procedure) within 15 mm proximal or distal to arteriotomy site based on pre-primary procedure CT angiography,
20. Target femoral artery diameter is less than 7 mm in diameter, based on pre-primary procedure CT angiography,
21. Further planned endovascular procedure in the target leg in the 30 days following the index procedure,
22. Subject is enrolled in another investigational medical device or drug study
23. Subject has been previously enrolled in this clinical study.
24. Current COVID-19 infection (with or without symptoms), recent positive test for COVID-19, or recent exposure (within two weeks) to a person with COVID-19 infection.

Procedural Exclusion Criteria If any Procedural Exclusion Criteria listed below, then closure with PerQseal®+ device is not permitted.

1. Initial common femoral arterial access achieved with manual palpation or blind arterial stick access, without use of an image guided approach (ultrasound or angiography).
2. Difficult dilation during initial target femoral artery access (e.g., that damages or kinks sheath dilators) while step-dilating up to the large-bore device,
3. During arterial puncture, the target femoral artery suspected to have experienced a back arterial wall needle puncture or underwent > one needle puncture during the primary procedure.
4. Subject has a tissue tract (i.e., estimated distance from skin entry point to arterial anterior surface at arteriotomy) expected to be greater than 8 cm,
5. Significant blood loss requiring transfusion of blood products during primary procedure or within 30 days prior to index procedure,
6. Activated clotting time (ACT) > 300 seconds immediately prior to sheath removal or if ACT measurements are expected to be > 300 seconds for more than 24 hours after index procedure,
7. Target puncture site is in a vascular graft,
8. Target arteriotomy greater than 26 F,
9. Target arteriotomy in the profunda femoris or superficial femoral artery or is in common femoral artery, but within 15 mm proximal of the bifurcation of the superficial femoral/ profunda femoris artery,
10. Target arteriotomy located at the level or above the inferior epigastric artery and/or beneath or above the inguinal ligament based on bony landmarks (above femoral head on A-P projection),
11. Subjects with an acute hematoma > 4 cm diameter, arteriovenous fistula, pseudoaneurysm, or intraluminal thrombosis at the target access site identified intra-procedurally,
12. Evidence of bleeding around the primary procedure sheath (BARC type 2 or higher),
13. Intra-procedural angiographic evidence of arterial laceration, dissection or stenosis within the femoral artery that would preclude use of the PerQseal®+ device,
14. Uncontrolled hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg) at the time of planned vascular closure,
15. Systolic blood pressure < 90 mmHg at the time of planned vascular closure.

    -

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Safety: Major Access Site Complications | though 30 days
  The primary safety endpoint is the rate of major access site complications attributable to the PerQseal® device. As per FDA definitions for Major access site complications.
Efficacy: Time to Haemostasis | 20 minutes
  Elapsed time in minutes from PerQseal® Introducer sheath removal to first observed cessation of common femoral artery (CFA) bleeding (excluding cutaneous or subcutaneous oozing, and in the absence of a developing hematoma).

SECONDARY OUTCOMES:
Safety: Incidence of Minor Access Site Complications | through 30 days
  Incidence and severity of minor access site complications attributable to the PerQseal® device, adapted from FDA-provided definitions.
Efficacy: PerQseal® Device Technical Success Rate | 10 minutes
  PerQseal® Device Technical Success Rate, defined as the number of PerQseal® devices that are deployed and achieve hemostasis (i.e., cessation of bleeding (excluding cutaneous or subcutaneous oozing)) without need for firm, adjunctive manual compression for greater than 10 minutes or alternative treatment (other than adjunctive endovascular ballooning) at target access site, divided by the total number of PerQseal® devices where deployment was attempted.
Efficacy: PerQseal® Treatment Success Rate | through 30 days
  PerQseal® Treatment Success Rate, defined as the number of subjects who meet PerQseal® Device Technical Success without experiencing a Major Access Site Complication, divided by the total number of subjects where PerQseal® device deployment was attempted.
Efficacy: Time to Device Deployment | 20 minutes
  Time to Device Deployment, defined as the time from insertion of the PerQseal® device into the PerQseal Introducer sheath to complete removal of the PerQseal® device delivery system and PerQseal® Introducer sheath from the subject following PerQseal® deployment.
Efficacy: Time to Ambulation | through 5 day
  Time to Ambulation is defined as: the elapsed time from PerQseal® + removal until the subject can walk 20 feet without re-bleeding at the target access site. This endpoint will be evaluated only for subjects who are ambulatory at the point of enrollment.
Efficacy: Total Closure Time | 40 minutes
  Total Closure Time is defined as: Time to Hemostasis (TTH) plus Time to Device Deployment

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - The Valley Hospital, Ridgewood, New Jersey
  - Weill Cornell Medicine, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Montefiore Hospital, The Bronx, New York
  - Lankenau Heart Institute, Wynnewood, Pennsylvania

IPD SHARING:
Plan to Share IPD: No